CLINICAL TRIAL: NCT07388420
Title: Adding Evolocumab to Conventional Lipid-lowering Therapy for Hypertriglyceridemia Induced Acute Pancreatitis: A Pilot Randomised Controlled Trial
Brief Title: Adding Evolocumab to Conventional Lipid-lowering Therapy for Hypertriglyceridemia Induced Acute Pancreatitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHNKKY-HTGAP
Record Dates: First submitted 2026-01-21; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Hypertriglyceridemia Induced Acute Pancreatitis
Keywords: Hypertriglyceridemia Induced Acute Pancreatitis; Evolocumab; Conventional lipid-lowering therapy
MeSH Terms: interventions — evolocumab; Fibric Acids; Heparin, Low-Molecular-Weight; Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional lipid-lowering therapy + Evolocumab group (Experimental)
  Interventions: Drug: Evolocumab 140 MG/ML [Repatha]
- Conventional lipid-lowering therapy group (Active Comparator)
  Interventions: Drug: Conventional lipid-lowering therapy

INTERVENTIONS:
Drug: Evolocumab 140 MG/ML [Repatha] — The clinicians strictly follow the treatment strategy for HTG-AP as stipulated in the 2021 "Emergency Expert Consensus on Diagnosis and Treatment of Hypertriglyceridemia Induced Acute Pancreatitis" to provide conventional lipid-lowering treatment for the patients, including dietary adjustments, fibrates, low-molecular-weight heparin, and insulin, etc. On the basis of conventional lipid-lowering treatment, 140mg of evolocumab is added by slow subcutaneous injection every two weeks, and the patients' responses are observed during this period.
  Other Names: Dietary adjustments; Fibrates; Low-molecular-weight heparin; Insulin
  Arms: Conventional lipid-lowering therapy + Evolocumab group
Drug: Conventional lipid-lowering therapy — This group only receives conventional lipid-lowering treatment without adding evolocumab.
  Other Names: Dietary adjustments; Fibrates; Low-molecular-weight heparin; Insulin
  Arms: Conventional lipid-lowering therapy group

SUMMARY:
The severity of hypertriglyceridemia induced acute pancreatitis (HTG-AP) is closely related to the serum triglyceride (TG) levels. The higher the TG levels, the greater the risk of developing severe acute pancreatitis (SAP). Previous expert consensus has pointed out that the key to treating HTG-AP is to rapidly lower serum TG levels to below 5.65 mmol/L. Evolocumab is a proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitor, which is often used to treat familial hypercholesterolemia, mixed dyslipidemia and atherosclerotic cardiovascular disease. At the same time, evolocumab also has the effect of reducing TG and may provide a feasible option for the management of HTG-AP. However, its efficacy and safety in reducing TG in patients with HTG-AP remain controversial. This study is a multicenter randomized controlled trial to evaluate the efficacy and safety of adding evolocumab to conventional lipid-lowering therapy in patients with HTG-AP.

DETAILED DESCRIPTION:
Overall, 40 patients with HTG-AP will be included. These patients will be randomly assigned in a 1:1 ratio to the conventional lipid-lowering therapy group and the conventional lipid-lowering therapy + evolocumab group. The primary endpoints are the TG levels at days 3 and 7 after treatment, and the rates of achieving TG levels below 5.65 mmol/L and 1.7 mmol/L at the same time points. Secondary endpoints include blood levels of total cholesterol (TC), high-density lipoprotein (HDL), low-density lipoprotein (LDL), and lipoprotein(a) at days 3 and 7; the incidence of recurrent acute pancreatitis (RAP), SAP, and other complications; as well as the length of hospital stay and total hospitalization costs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18~75 years
* Patients with HTG-AP
* Mixed hyperlipidemia
* Sign the informed consent form

Exclusion Criteria:

* Patients who have received lipid-lowering drugs or blood purification treatment
* Patients who have used evolocumab within one month before admission
* Patients who are accompanied by diseases that can seriously affect the survival
* Patients who have participated in the clinical research of other drugs within one month
* Patients who are pregnant or breastfeeding
* Patients with allergic asthma, allergic urticaria, eczema, and those who have a clear history of multiple drug and food allergies
* Other circumstances that researchers consider not suitable for participation in this study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The TG levels on the 3rd and 7th days after treatment | 3 days and 7days
The rates of achieving TG levels below 5.65 mmol/L and 1.7 mmol/L on the 3rd and 7th days after treatment | 3 days and 7 days

SECONDARY OUTCOMES:
The serum levels of TC, HDL, LDL, and lipoprotein(a) on the 3rd and 7th days after treatment | 3 days and 7days
The incidence of RAP, SAP, and other complications | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zengwu Wang, Jing Liu, Jianjun Li, et al. Chinese Guidelines for Lipid Management (2023). Chinese Journal of Circulation. 2023; 38 (03) : 237-271.
- [Background] Wu BU, Johannes RS, Sun X, Tabak Y, Conwell DL, Banks PA. The early prediction of mortality in acute pancreatitis: a large population-based study. Gut. 2008 Dec;57(12):1698-703. doi: 10.1136/gut.2008.152702. Epub 2008 Jun 2. PMID 18519429
- [Background] Ong Y, Shelat VG. Ranson score to stratify severity in Acute Pancreatitis remains valid - Old is gold. Expert Rev Gastroenterol Hepatol. 2021 Aug;15(8):865-877. doi: 10.1080/17474124.2021.1924058. Epub 2021 May 13. PMID 33944648
- [Background] Banks PA, Bollen TL, Dervenis C, Gooszen HG, Johnson CD, Sarr MG, Tsiotos GG, Vege SS; Acute Pancreatitis Classification Working Group. Classification of acute pancreatitis--2012: revision of the Atlanta classification and definitions by international consensus. Gut. 2013 Jan;62(1):102-11. doi: 10.1136/gutjnl-2012-302779. Epub 2012 Oct 25. PMID 23100216
- [Background] Qi R, Liu H, Li X, Chen M. Successful use of Proprotein Convertase Subtilisin/Kexin Type 9 Inhibitors in Hypertriglyceridemia-induced Acute Pancreatitis: A Case Report. Curr Cardiol Rev. 2025;21(3):e1573403X343784. doi: 10.2174/011573403X343784241115055037. PMID 39773061
- [Background] Chen H, Li X, Chen J, Zhao Y, Zhang W, Li H, Qi X. Lipid-lowering effect of evolocumab in hypertriglyceridemia-induced acute pancreatitis. Eur J Pharmacol. 2025 Nov 5;1006:178148. doi: 10.1016/j.ejphar.2025.178148. Epub 2025 Sep 16. PMID 40967356
- [Background] Lu W, Wang L, Du C, Qin L, Li J, Wang H. PCSK9 Inhibitors in Multi-Branch Lesions in Coronary Artery Disease with Substandard Lipid-Lowering Effects. Altern Ther Health Med. 2024 Aug;30(8):356-360. PMID 38064616
- [Background] Raal FJ, Stein EA, Dufour R, Turner T, Civeira F, Burgess L, Langslet G, Scott R, Olsson AG, Sullivan D, Hovingh GK, Cariou B, Gouni-Berthold I, Somaratne R, Bridges I, Scott R, Wasserman SM, Gaudet D; RUTHERFORD-2 Investigators. PCSK9 inhibition with evolocumab (AMG 145) in heterozygous familial hypercholesterolaemia (RUTHERFORD-2): a randomised, double-blind, placebo-controlled trial. Lancet. 2015 Jan 24;385(9965):331-40. doi: 10.1016/S0140-6736(14)61399-4. Epub 2014 Oct 1. PMID 25282519
- [Background] Blom DJ, Hala T, Bolognese M, Lillestol MJ, Toth PD, Burgess L, Ceska R, Roth E, Koren MJ, Ballantyne CM, Monsalvo ML, Tsirtsonis K, Kim JB, Scott R, Wasserman SM, Stein EA; DESCARTES Investigators. A 52-week placebo-controlled trial of evolocumab in hyperlipidemia. N Engl J Med. 2014 May 8;370(19):1809-19. doi: 10.1056/NEJMoa1316222. Epub 2014 Mar 29. PMID 24678979
- [Background] Tan H, Li W, Huang Z, Han Y, Huang X, Li D, Xing X, Monsalvo ML, Wu Y, Mao J, Xin L, Chen J; HUA TUO study investigators. Efficacy and Safety of Evolocumab in Chinese Patients with Primary Hypercholesterolemia and Mixed Dyslipidemia: 12-Week Primary Results of the HUA TUO Randomized Clinical Trial. Cardiol Ther. 2023 Jun;12(2):341-359. doi: 10.1007/s40119-023-00304-x. Epub 2023 Feb 21. PMID 36802321
- [Background] Wiggins BS, Senfield J, Kassahun H, Lira A, Somaratne R. Evolocumab: Considerations for the Management of Hyperlipidemia. Curr Atheroscler Rep. 2018 Mar 6;20(4):17. doi: 10.1007/s11883-018-0720-3. PMID 29511875
- [Background] Lu Z, Zhang G, Guo F, Li M, Ding Y, Zheng H, Wang D. Elevated triglycerides on admission positively correlate with the severity of hypertriglyceridaemic pancreatitis. Int J Clin Pract. 2020 Mar;74(3):e13458. doi: 10.1111/ijcp.13458. Epub 2019 Dec 14. PMID 31799779
- [Background] Xin Hong, Liming Wang, Zhengliang Zhang, et al. Emergency Expert Consensus on Diagnosis and Treatment of Hypertriglyceridemia Induced Acute Pancreatitis [J]. Chinese General Practice, 2021, 24(30): 3781-93
- [Background] Na Zhang, Haiyan Zhang, Xiaohong Guo, et al. Meta-analysis of etiological changes of acute pancreatitis in China in the past Decade [J]. Chinese Journal of Gastroenterology and Imaging (Electronic Edition), 2016, 6(02): 71-5
- [Background] Pancreatic Surgery Group, Surgical Branch of the Chinese Medical Association Chinese Guidelines for Diagnosis and Treatment of Acute Pancreatitis (2021) [J]. Chinese Journal of Digestive Surgery, 2021, 20(07): 730-9.